CLINICAL TRIAL: NCT04644458
Title: Use of Ulna Length to Predict Protective Lung Tidal Volume in Adult Egyptians
Brief Title: Use of Ulna Length to Predict Tidal Volume in Adult Egyptians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Bahaa Mohammed Refaie, Lecturer of anesthesia and ICU, Sohag University
Other Study IDs: 1990
Record Dates: First submitted 2020-11-15; First posted 2020-11-25 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Tidal Volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measuring the ulna length using meauring tape — the left ulna will be measured with a measure tape from the olecranon to mid point of styloid process.

SUMMARY:
The aim of the study is to evaluate the ability of ulna length to predict accurate protective lung tidal volume in Egyptian people in reference to their standing height.

DETAILED DESCRIPTION:
After approval of local ethical committee and informed consent, one hundred healthy volunteers will be rnrolled in this study. Height of each subject will be measured while standing upright against a wall. Then, the left ulna will be measured with a measure tape from the olecranon to mid point of styloid process. From ulna length, height is estimated as advised by Malnutrition Advisory Group, British Association of Parenteral and Enteral Nutrition. October 2008. Malnutrition Universal Screening Tool.Protective lung tidal volume is calculated as 6 ml/kg predicted body weight (PBW) as follow:

PBW= 50*0.91 (centimetres of height - 152.4) in males and 45.5*0.91(centimetres of height - 152.4) in females.

Each measurement will be performed only once for each subject. Agreement between measurements will be expressed by the Bland-Altman method.

ELIGIBILITY:
Inclusion Criteria:

- Healthy adult Egyptian

Exclusion Criteria:

- Deformity or previous surgery in the left arm

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Adult Egyptian volunteers
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Protective lung tidal volume | measurement of left ulna while standing for each volunteer throught the study completion, average 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hosam eldeen M Marie, MD, Study Director — Consultant of anesthesia and ICU Elhelal insurance hospital
Locations (1):
- Sohag university hospital, Sohag, Egypt